CLINICAL TRIAL: NCT00390026
Title: A Prospective, Randomized, Double-masked, Controlled Study on Intravitreal Bevacizumab (Avastin) Versus Verteporfin (Visudyne) Photodynamic Therapy (PDT) for Patients With Neovascular Age-related Macular Degeneration (AMD)
Brief Title: The Avastin vs Visudyne for Neovascular AMD Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lucentis, a treatment superior to PDT, has become available i Sweden.
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Anders Kvanta, Professor, St. Erik Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVA001; EU2006-001200-36
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Age-related Macular Degeneration
Keywords: Neovascular age-related macular degeneration; Bevacizumab; Photodynamic therapy
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

ARMS (2):
- Avastin (Experimental)
  Interventions: Drug: Bevacizumab (Avastin); Drug: Verteporfin photodynamic therapy (PDT)
- Visudyne (Active Comparator)
  Interventions: Drug: Bevacizumab (Avastin); Drug: Verteporfin photodynamic therapy (PDT)

INTERVENTIONS:
Drug: Bevacizumab (Avastin)
Drug: Verteporfin photodynamic therapy (PDT)

SUMMARY:
The object of the study is to compare the treatment effect of bevacizumab (Avastin), an antibody targeting vascular endothelial growth factor, with verteporfin photodynamic therapy (PDT) for patients with neovascular age-related macular degeneration, the leading cause of vision severe loss in the Western world.

DETAILED DESCRIPTION:
Neovascular age-related macular degeneration (AMD) is caused by an ingrowth of pathological vessels under the macula. Experimental studies have demonstrated that vascular endothelial growth factor (VEGF) is centrally involved in this process. Current treatment options have up until now been limited to photodynamic therapy (PDT) where a photosensitizing agent in combination with laser is used to occlude the pathologic vessels. Anti-VEGF agents have recently become available making them a potentially attractive treatment alternative for neovascular AMD. We will compare the effect intravitreally administered bevacizumab with conventional PDT in a prospective, randomized and controlled trial including 100 patients (50 patients receiving either treatment regimen). Non-treated patients will receive either sham-injection or sham-PDT. The primary endpoint of the study is the amount of patients losing less than 15 letters on the ETDRS visual acuity chart. The study will go on for 2 years with an interim report after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* patients with subfoveal neovascular AMD with either classic/predominantly classic or small occult lesions
* visual acuity >=0.1

Exclusion Criteria:

* patients with subfoveal neovascular AMD with minimally classic lesions or large occult lesions
* subfoveal hemorrhage (>1DA) or fibrosis
* patients previously treated for neovascular AMD in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients losing less than 15 letters on the ETDRS visual acuity chart. | 1 year

SECONDARY OUTCOMES:
Proportion of patients gaining more than 15 letters on the ETDRS visual acuity chart. | 1 year
Proportion of patients losing more than 30 letters on the ETDRS visual acuity chart. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kvanta, MD, PhD, Principal Investigator — S:t Erik's Eye Hospital; Stefan Seregard, MD, PhD, Study Director — S:t Eriks Eye Hospital
Locations (1):
- S:t Eriks Eye Hospital, Stockholm, Sweden

REFERENCES:
- See also: Hospital homepage — http://www.sankterik.se